CLINICAL TRIAL: NCT03221569
Title: Ketamine v. Ketorolac for Management of Generalized Tension Type Headache
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Brooklyn Hospital Center (Other)
Responsible Party: Principal Investigator, Billy Sin, Director, Emergency Medicine Clinical Research Program, The Brooklyn Hospital Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 779354-2
Record Dates: First submitted 2017-07-17; First posted 2017-07-18 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Ketorolac; Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Arm A would include 0.3mg/kg intravenous piggyback ketamine and 1cc normal saline as placebo via intravenous push while Arm B would receive 50ml normal saline and ketorolac 30mg.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Aside from primary investigator (B.Sin) and pharmacist procuring the study interventions, blinding will be applied to patient, physicians, nurses, research associates responsible for collect data and also the independent biostatistician responsible for evaluating the data. Patients will be randomized to receive study numbers that corresponds to treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intravenous ketamine (Experimental): Arm will include 0.3 mg/kg intravenous piggyback ketamine over 10 minutes for 1 dose and a 1ml normal saline placebo via intravenous push
  Interventions: Drug: Intravenous ketamine; Drug: Normal saline
- ketorolac (Active Comparator): Arm will include 30mg ketorolac intravenous push and 50ml normal saline over 10 minutes
  Interventions: Drug: Ketorolac; Drug: Normal saline

INTERVENTIONS:
Drug: Intravenous ketamine — 0.3mg/kg IVPB over 15 minutes
  Other Names: ketamine intravenous
  Arms: Intravenous ketamine
Drug: Ketorolac — as active comparator, will be administered together with metoclopramide in one normal saline 50ml bag
  Arms: ketorolac
Drug: Normal saline — Will be given as 50ml intravenous bag as placebo for double-blinding purposes in patients who will also receive intranasal ketamine.
  Will be prepared in intranasal syringe for double blinding purposes for patients who are randomized to receive intranasal ketamine.
  Other Names: saline
  Arms: Intravenous ketamine
Drug: Normal saline — 1ml intravenous push as placebo for double-blinding purposes
  Other Names: saline
  Arms: ketorolac

SUMMARY:
The hypothesis of the study is that sub-dissociative dose ketamine will prove to be superior to or as standard therapy, ketorolac, in the treatment of acute tension type headache (TTH) as measured by the 10 point Numerical Rating Scale (NRS. The aim of the study is to compare the safety & efficacy of intravenous sub-dissociative dose ketamine versus ketorolac for acute treatment of migraines in the Emergency Department (ED) The primary endpoints are: Patient perception of pain as described by the use the Numerical Rating Scale (NRS) at 30 minutes.

The secondary endpoints are: Frequency and mean dose of rescue/additional doses of therapy at 15, 30, 45, 60, 75, 90 min, Number of emergency department re-visits for acute migraine one month post discharge, incidence of dissociative effects (characterized by hallucination, disorientation, confusion, agitation, delirium, dreams) during study period, incidence of nausea, vomiting, or worsening headache, Incidence of bad taste, Incidence of burning sensations in the nostrils, incidence of hypertension, time to patient discharge from the initiation of study medication/placebo, patient satisfaction of pain control based on a Likert Scale.

DETAILED DESCRIPTION:
This will be a "double-dummy" study in that there will be no placebo only arm. Medications will be administered in a double blind randomized fashion. Patients would be enrolled in Arm A or Arm B depending upon the initial randomization. Arm A would include 0.3 mg/kg ketamine into a 100 cc normal saline IV bag and normal saline injection (1ml) while Arm B would receive 100cc of normal saline and 30mg of ketorolac intravenously.

An order would be placed by the medical resident, medical attending, a study investigator who is a physician, or a pharmacist under the permission of the attending physician into Allscripts for a study intervention. Upon receiving the order in Allscripts, the order would be verified by the pharmacy. All medications will be prepared in pharmacy, which will maintain a master list of contents of each sealed envelope. Once notified of which envelope has been pulled, the pharmacist will prepare either arm. ED personnel will obtain the infusion preparation from pharmacy. It will be labeled for the patient, with study number, but without other identifying marks. When the study medication is picked up, pharmacy will open the sealed envelope to confirm which medication arm was prepared in order to internally verify the correct preparation. The nurse assigned to the patient would administer the intervention. A research associate or a study investigator would approach the patient to assess and record primary outcomes, secondary outcomes at designed time intervals. The data will be recorded on the data collection instrument. If additional medication is requested by the patient, the orders would be placed by the medical resident or attending who are assigned to the patient in the ED. Upon completion of the treatment portion of the study, patients will be asked of the participant's satisfaction with therapy. Only the patient who signed the consent form will be allowed to answer the questions.

All data retrieved from the paper data collection sheets will be transcribed into an encrypted and password protected electronic database by the research associate. All patient identifiers would be de-identified in the database. All participants would be assigned a study participant number.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are: Patients 18-65 years old who provides informed consent and presents to the ED with an acute tension type headache (TTH), as classified by meeting the following:

  1. Have at least 10 episodes of headache occurring on average less than 12 days per year AND Fullfuling B-D B. Lasting 30mins to 7 days C. At least 2 of the following 4 criteria

  <!-- -->

  1. bilateral location
  2. pressing/tightening (non-pulsating)
  3. mild or moderate
  4. not aggravated by routine physical activity such as walking or climbing stairs D. Both of the following

  <!-- -->

  1. no nausea/vomiting
  2. No more than one of photophobia or phonophobia

Exclusion Criteria: Non migraine primary headache disorder or unclassifiable, previous enrollment in study, fever >100.3, Patients with suspected secondary headache disorder such as SAH or sinusitis, performance of lumbar puncture or potential need for LP, Severe hypertension (≥180/100), History of CAD or hypertension, presence of/suspected for traumatic head injury in the past 30 days with or without loss of consciousness, Presence of/suspected for myocardial ischemia, presence of/suspected for alcohol intoxication, Hemodynamic instability, history of psychiatric disorders, known or suspected pregnancy or breast feeding, allergy to ketamine, ketorolac, previous enrollment in the study, patients with language barriers, refusal to provide consent to receive intravenous therapy, reported illicit drug use within the past 5 days, patients weighing over 100kg

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Pain scores | At 30 minutes after initiation of study intervention
  10 point number rating scale

SECONDARY OUTCOMES:
Incidence of adverse events | throughout study period (105 mins)
  adverse events reported in each group
mean dose of rescue analgesia required | throughout study period (105 minutess)
  dose of rescue analgesia required in each group
length of stay | throughout study period (105 minutes)
  median ED length of stay in each group

CONTACTS AND LOCATIONS:
Locations (1):
- The Brooklyn Hospital Center, Brooklyn, New York, United States